CLINICAL TRIAL: NCT04731103
Title: Inhibition of Reverse Transcription in Type I Interferon Mediated Neuropathology
Brief Title: Inhibition of Reverse Transcription in Aicardi-Goutières Syndrome
Acronym: AGS-RTI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AC19167
Record Dates: First submitted 2020-07-14; First posted 2021-01-29 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-06

CONDITIONS: Aicardi-Goutières Syndrome
Keywords: Type 1 Interferon; Reverse Transcriptase Inhibitor(s)
MeSH Terms: interventions — abacavir; Lamivudine

STUDY DESIGN:
Intervention Model Description: Open label, non-placebo controlled. We propose a trial design involving an initial no-drug period of six weeks followed by three treatment arms each of six weeks, with a washout period of four weeks between treatment arms (considering documented drug half-lives).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abacavir (ABC) (Active Comparator): Participants receive Abacavir (ABC) for 6 weeks and 4 weeks of washout.
  Interventions: Drug: Abacavir (ABC)
- Lamivudine (3TC) (Active Comparator): Participants receive Lamivudine (3TC) for 6 weeks and 4 weeks of washout.
  Interventions: Drug: Lamivudine (3TC)
- Abacavir (ABC)+Lamivudine (3TC)+Zidovudine (AZT) (Active Comparator): Participants receive Abacavir (ABC)+Lamivudine (3TC)+Zidovudine (AZT) for 6 weeks and 4 weeks of washout.
  Interventions: Drug: Abacavir (ABC)+Lamivudine (3TC)+Zidovudine (AZT)

INTERVENTIONS:
Drug: Abacavir (ABC) — Tablets or oral solution
  Arms: Abacavir (ABC)
Drug: Lamivudine (3TC) — Tablet or oral solution
  Arms: Lamivudine (3TC)
Drug: Abacavir (ABC)+Lamivudine (3TC)+Zidovudine (AZT) — Tablet or oral solution
  Arms: Abacavir (ABC)+Lamivudine (3TC)+Zidovudine (AZT)

SUMMARY:
Aicardi-Goutières syndrome (AGS) is a disease of children, particularly affecting the brain and the skin. There is a close link between AGS and increased amounts of a chemical called interferon. Normally humans only produce interferon when they are infected with a virus. In AGS, there is no viral infection. Instead, the cells in the cells of affected patients are confused into thinking that their own genetic material is coming from a virus. As a result they produce interferon all the time, which acts as a poison that damages the cells. The Investigators wish to treat AGS patients with drugs called reverse transcriptase inhibitors (RTIs), used to fight the HIV-1 virus that causes AIDS. The investigators will monitor the effect of treatment on interferon levels, and look at other markers which might give us clues to how the drugs are working. The trial is funded by the Medical Research Council, and involves experts based in Edinburgh, Birmingham, Manchester and Great Ormond Street Hospital.

DETAILED DESCRIPTION:
Aicardi-Goutières syndrome (AGS) is a severe childhood disease of the brain associated with very high levels of a chemical called type I interferon. Normally humans only produce interferon when they are infected with a virus. In AGS, there is no obvious viral infection. Instead, due to changes (mutations) in the genetic code in these individuals, it is believed that the cells in the body are fooled into thinking that the person's own DNA is viral - that is to say, there is a confusion in telling 'self' from 'non-self'.

In fact, a large amount of our own DNA is made up of ancient virus (called 'endogenous retrovirus' and sometimes also referred to as 'junk DNA'), that have been included into our own genetic material over millions of years. These endogenous retroviruses can still act like a virus coming from outside of the body, so that they need to be controlled. The Investigators have wondered if the genetic changes causing AGS mean that these normal control mechanisms don't work. If that is true, the endogenous retroviruses could start to make copies of themselves which might be recognised by our immune system as 'non-self' ('foreign' i.e. viral), leading to the continuous production of interferon which then damages the cells in our body.

Since humans cannot repair the genetic code in every cell, the investigators wish to treat AGS patients with drugs called reverse transcriptase inhibitors (RTIs). RTIs are used to fight the HIV-1 virus that causes AIDS. In the case of AGS, it is not treating HIV-1, but the investigators wonder if the same drugs might be able to control endogenous retroviruses that are driving interferon production. Indeed, in a recently completed study the investigators gathered early information to suggest that treatment of patients with AGS with RTIs for one year did lead to a reduction in interferon, with levels increasing again when we stopped the drugs.

The current study will involve three treatment arms, and an assessment of interferon status and other markers which we think will give us information about AGS, and about how RTIs may work in the treatment of AGS.

This study is of potential importance for patients with AGS and their families since there are no licenced drugs for this disorder at the present time. Scientifically, the project will be of considerable interest if the results support the possibility that 'junk DNA' can be associated with human disease. RTIs are very safe drugs, that have been used in millions of people with HIV-1 around the world. If the results turn out to be convincing, the investigators believe that it might be worth thinking about using RTIs to treat other diseases that have also been linked to increased levels of type I interferon, for example the relatively common immune condition called systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mutations in any of TREX1, the three components of the RNase H2 complex (RNASEH2A, RNASEH2B, RNASEH2C: considered as one genotype) or SAMHD1.
* Greater than age 3 months and less than 16 years of age at the time of recruitment
* Resident in the United Kingdom (UK)
* Informed Consent obtained from parent or personal legal representative
* For inclusion in the study, a patient has either to have completed the vaccination programme two weeks prior to starting the trial, or remain unvaccinated until the end of the trial, or agree to defer vaccination until immediately after a study drug arm, so that there is a period of at least two weeks following vaccination and before the start of the following drug arm.

Exclusion Criteria:

* Patients with AGS due to mutations in ADAR1 and IFIH1 will not be considered, given that the induction of interferon relating to these genotypes does not involve a reverse transcription step.
* Pre-existing disease, not due to AGS, which would preclude the use of zidovudine, lamivudine and abacavir
* Patients with abnormally low neutrophil counts (<0.75 x 109/l) and / or abnormally low haemoglobin levels (<7.5 g/dl)(particularly relevant to zidovudine), significant renal (creatinine clearance < 50 ml/min; particularly relevant to lamivudine) or significant hepatic impairment (particularly relevant to abacavir; avoid if Child Pugh > 5)
* Participation in another Clinical Trial of an Investigational Medicinal Product (CTIMP) trial
* Pregnancy
* Breast feeding
* Hepatitis B and C infection
* Potential hypersensitivity to abacavir, assessed according to HLA-B*5701 status
* Hypersensitivity to the active substances or to any of the excipients listed in section 6.1 of the Summary of Product Characteristics (SPC)
* Where, in the opinion of the Investigator the participant cannot fulfil the requirements of the trial protocol

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Determine if the use of the reverse transcriptase inhibitors abacavir (ABC), lamivudine (3TC) and zidovudine (AZT) reduces Interferon (IFN) signalling in patients with mutations in TREX1, RNASEH2A, RNASEH2B, RNASEH2C or SAMHD1 | At 6 weeks
  The primary outcome is a change in the Interferon(IFN) score over baseline at 6 weeks end of treatment.

SECONDARY OUTCOMES:
A change in interferon alpha protein levels | 6 weeks
  Change in interferon alpha protein levels (fg/ml) over 6 weeks per treatment arm.
A change in cerebral blood flow | 6 weeks
  Change in cerebral blood flow (ml/min/100g of tissue) over 6 weeks per treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Yanick Crow, Principal Investigator — University of Edinburgh
Locations (1):
- Yanick Crow, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rice GI, Meyzer C, Bouazza N, Hully M, Boddaert N, Semeraro M, Zeef LAH, Rozenberg F, Bondet V, Duffy D, Llibre A, Baek J, Sambe MN, Henry E, Jolaine V, Barnerias C, Barth M, Belot A, Cances C, Debray FG, Doummar D, Fremond ML, Kitabayashi N, Lepelley A, Levrat V, Melki I, Meyer P, Nougues MC, Renaldo F, Rodero MP, Rodriguez D, Roubertie A, Seabra L, Uggenti C, Abdoul H, Treluyer JM, Desguerre I, Blanche S, Crow YJ. Reverse-Transcriptase Inhibitors in the Aicardi-Goutieres Syndrome. N Engl J Med. 2018 Dec 6;379(23):2275-7. doi: 10.1056/NEJMc1810983. No abstract available. PMID 30566312